CLINICAL TRIAL: NCT01468441
Title: Effect of Ovarian Stimulation Using Recombinant FSH and GHRH Antagonist in Alternate Days on ICSI Outcomes
Brief Title: Ovarian Stimulation Using Recombinant Follicle-stimulating Hormone (FSH) and Gonadotrophin Releasing Hormone (GnRH) Agonist in Alternate Days
Acronym: Gonapeptyl
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fertility - Assisted Fertilization Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Fert-LG-Doutorado
Record Dates: First submitted 2011-10-31; First posted 2011-11-09 (Estimated); Last update posted 2012-07-13 (Estimated); Status verified 2012-07

CONDITIONS: Infertility
Keywords: ovarian stimulation; GnRH agonist; GnRH antagonist; hCG microdose; ICSI
MeSH Terms: conditions — Infertility | interventions — Triptorelin Pamoate; cetrorelix

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- GnRH agonist (Experimental): Administration of GnRH agonist in alternate days, recombinant FSH and hCG microdose for ovarian stimulation.
  Interventions: Drug: Triptorelin
- GnRH antagonist (Active Comparator): Daily administration of GnRH antagonist, recombinant FSH and hCG microdose for ovarian stimulation.
  Interventions: Drug: Cetrorelix

INTERVENTIONS:
Drug: Triptorelin — Triptorelin (0.1 mg, Gonapeptyl® Daily; Ferring, Kiel, Germany) in alternate-days from Day 1 of the menstrual cycle until the day of hCG administration.
  Other Names: Gonapeptyl
  Arms: GnRH agonist
Drug: Cetrorelix — When patients presented at least two follicles ≥ 14mm upon scan on days 7- 9, GnRH antagonist (cetrorelix, 0.25 mg/day, Cetrotide®; EMD Serono, Inc, Rockland, MA, USA) administration is started and continued until hCG administration.
  Other Names: Cetrotide
  Arms: GnRH antagonist

SUMMARY:
The present prospective study was designed to compare the effects of administering a daily dose of gonadotrophin releasing hormone (GnRH) antagonist vs. an alternate-day dosage of GnRH agonist on ovarian response and in vitro fertilization (IVF) outcome in patients stimulated with recombinant follicle-stimulating hormone (FSH) and human chorionic gonadotrophin (hCG) microdose.

DETAILED DESCRIPTION:
Inclusion criteria were as follows: women of good physical and mental health, under 37 years old, with regular menstrual cycles of 25-35 days, normal basal FSH and luteinizing hormone (LH) levels, body mass index (BMI) less than 30 kg/m2, presence of both ovaries and intact uterus, absence of polycystic ovaries, endometriosis, or gynaecological / medical disorders and a negative result in a screening for sexually transmitted diseases.

No patient had received any hormone therapy for at least 60 days preceding the study. Eligible patients who agreed to participate were randomized in two treatment groups. Patients were allocated to a GnRH analogue treatment group according to a computer-generated randomization table.

ELIGIBILITY:
Inclusion Criteria:

* women of good physical and mental health
* under 37 years old, with regular menstrual cycles of 25-35 days
* normal basal FSH and LH levels
* BMI less than 30 kg/m2
* presence of both ovaries and intact uterus
* absence of polycystic ovaries
* endometriosis, or gynaecological / medical disorders and a negative result in a screening for sexually transmitted diseases
* all patients signed a written informed consent form
* no patient had received any hormone therapy for at least 60 days preceding the study.

Max Age: 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 96 (Actual)
Dates: Start 2011-09; Primary Completion 2012-03 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
cost of treatment | One month

SECONDARY OUTCOMES:
Implantation and pregnancy rates | 2 months

CONTACTS AND LOCATIONS:
Overall Officials: Luiz Guilherme Maldonado, M.Sc., Principal Investigator — Fertility - Assisted Fertilization Center
Locations (1):
- Fertility - Assisted Fertilization Center, São Paulo, São Paulo, Brazil

REFERENCES:
- [Derived] Maldonado LG, Franco JG Jr, Setti AS, Iaconelli A Jr, Borges E Jr. Cost-effectiveness comparison between pituitary down-regulation with a gonadotropin-releasing hormone agonist short regimen on alternate days and an antagonist protocol for assisted fertilization treatments. Fertil Steril. 2013 May;99(6):1615-22. doi: 10.1016/j.fertnstert.2013.01.095. Epub 2013 Feb 5. PMID 23394779